CLINICAL TRIAL: NCT03441945
Title: New Method: Can Magnetic Steering Enhance Capsule Gastroscopy Gastric Emptying?
Brief Title: Magnetic Steering Enhance Capsule Gastroscopy Gastric Emptying
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhuan Liao (Other)
Responsible Party: Sponsor-Investigator, Zhuan Liao, professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MS-enhance-MCCG-GE
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Capsule Endoscopy; Gastric Emptying
Keywords: Magnetic; Capsule Endoscopy; enhance; gastric emptying

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): The patients swallowed the capsule with water in the lying position.After finishing the stomach examination, the operation of the capsule is adjusted to "small bowel mode" without magnetic control. Capsule entered the duodenum under physiological peristalsis. The position of the capsule was established using a real-time viewer. If the capsule failed to enter the duodenum after one hour, domperidone (10 mg) was orally administered.
- magnetic steering (Experimental): After finishing the stomach examination as the control protocol, the capsule was lifted with the magnetic control, then rotating the capsule until the camera end oriented toward the pylorus . Next, the endoscopist could drag the capsule close to the pylorus with the guidance magnet robot, waiting for the open of pylorus. Once the pylorus opened, the capsule could enter the duodenum with gastric peristalsis. After reaching the duodenal bulb, capsule was held to the maximum position of "Z", then the capsule would scan the duodenal bulb automatically with the mode "360° automatic scanning".
  Interventions: Other: magnetic steering

INTERVENTIONS:
Other: magnetic steering — magnetic steering
  Arms: magnetic steering

SUMMARY:
The research continuously enrolled 100 patients undergone MCCG between May to December 2017 as the intervention group with magnetic steering of capsule in the pylorus and duodenum, and randomly selected 100 patients before May 2017 from the database as the control group with passive movement of the capsule. The difference of the pyloric transit time (PTT) and duodenal papilla detection rate (DPDR) between the two groups were compared, and related factors were also investigated.

DETAILED DESCRIPTION:
Background and Aims: Capsule endoscopy is a valuable tool in the diagnosis of small bowel disease. However, the incompletion of small bowel examination may reduce the diagnostic accuracy, which mainly caused by delayed capsule gastric emptying. Thus the aim of this study was to validate the effect of magnetic steering on enhancing gastric emptying and mucosal visualization within duodenum during magnetically controlled capsule gastroscopy (MCCG) examination.

Methods: As a historical prospective cohort study, the research continuously enrolled 100 patients undergone MCCG between May to December 2017 as the intervention group with magnetic steering of capsule in the pylorus and duodenum, and randomly selected 100 patients before May 2017 from the database as the control group with passive movement of the capsule. The difference of the pyloric transit time (PTT) and duodenal papilla detection rate (DPDR) between the two groups were compared, and related factors were also investigated.

ELIGIBILITY:
Inclusion Criteria:

1. patients over 18 years of age undergone MCCG examination in Changhai Hospital

Exclusion Criteria:

1. pregnancy or suspected pregnancy;
2. suspected or known intestinal stenosis;
3. pacemaker, other implanted electro medical devices which could interfere with magnetic resonance; (4) undergone a known surgery which could possibly affect visualization of the duodenal papilla;

(5) other conditions which may lead to capsule retention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
PTT | 3 month
  pyloric transit time

SECONDARY OUTCOMES:
DPDR | 3 month
  duodenal papilla detection rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
We may share IPD when we finish this study

REFERENCES:
- [Background] Zou WB, Hou XH, Xin L, Liu J, Bo LM, Yu GY, Liao Z, Li ZS. Magnetic-controlled capsule endoscopy vs. gastroscopy for gastric diseases: a two-center self-controlled comparative trial. Endoscopy. 2015 Jun;47(6):525-8. doi: 10.1055/s-0034-1391123. Epub 2015 Jan 15. PMID 25590177
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Lee MM, Jacques A, Lam E, Kwok R, Lakzadeh P, Sandhar A, Segal B, Svarta S, Law J, Enns R. Factors associated with incomplete small bowel capsule endoscopy studies. World J Gastroenterol. 2010 Nov 14;16(42):5329-33. doi: 10.3748/wjg.v16.i42.5329. PMID 21072896
- [Background] Clarke JO, Giday SA, Magno P, Shin EJ, Buscaglia JM, Jagannath SB, Mullin GE. How good is capsule endoscopy for detection of periampullary lesions? Results of a tertiary-referral center. Gastrointest Endosc. 2008 Aug;68(2):267-72. doi: 10.1016/j.gie.2007.11.055. Epub 2008 Apr 18. PMID 18378233
- [Result] Hale MF, Drew K, Sidhu R, McAlindon ME. Does magnetically assisted capsule endoscopy improve small bowel capsule endoscopy completion rate? A randomised controlled trial. Endosc Int Open. 2016 Feb;4(2):E215-21. doi: 10.1055/s-0035-1569846. PMID 26878053
- [Derived] Jiang X, Qian YY, Liu X, Pan J, Zou WB, Zhou W, Luo YY, Chen YZ, Li ZS, Liao Z. Impact of magnetic steering on gastric transit time of a capsule endoscopy (with video). Gastrointest Endosc. 2018 Oct;88(4):746-754. doi: 10.1016/j.gie.2018.06.031. Epub 2018 Jul 11. PMID 30005825